CLINICAL TRIAL: NCT00529555
Title: A 9 Month,3-arm Multicenter Clinical Trial of Treatment With Periocline Gel (2.1% Minocycline HCl) for Adjunctive Use to Scaling and Root Planing (SRP) in Adults With Periodontal Disease.
Brief Title: Periocline as an Adjunct to Scaling and Root Planing for Adult Periodontitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunstar Americas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SB-PER-05-001
Record Dates: First submitted 2007-09-11; First posted 2007-09-14 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Adult Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Scaling and root planing + SHAM TX (Sham Comparator): sham treatment
  Interventions: Procedure: Scaling and root planing
- Scaling and root planing + Vehicle (Placebo Comparator): Placebo
  Interventions: Procedure: Scaling and root planing
- Scaling & root planing + Periocline Gel (Active Comparator): Minocycline HCL 2.1%
  Interventions: Drug: minocycline HCl 2.1%

INTERVENTIONS:
Drug: minocycline HCl 2.1% — Minocycline HCl 2.1% gel as an adjunct to scaling and root planing. Dosing is by topical delivery into gingival pockets at baseline, 2 weeks, 4 weeks, 3 months and 6 months.
  Other Names: periocline
  Arms: Scaling & root planing + Periocline Gel
Procedure: Scaling and root planing — scaling and root planing
  Other Names: SRP
  Arms: Scaling and root planing + SHAM TX; Scaling and root planing + Vehicle

SUMMARY:
Periodontal disease (commonly called gum disease) is generally treated by deep cleaning of the root surfaces of the teeth. This is also called scaling and root planing. Placing a topical antibiotic into the periodontal pocket at the time of scaling and root planing may help reduce pocket depth and thus help the periodontal disease. Periocline (minocycline HCl) 2.1% gel is a topical antibiotic approved in a number of countries for this use, and is now being tested in the US.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe periodontitis

Exclusion Criteria:

* recent periodontal therapy
* certain medical or dental conditions
* pregnancy
* allergy to active drug or related drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Genco, DDS, PhD, Principal Investigator — State University of New York at Buffalo
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - San Francisco, San Francisco, California
  - University of Florida, Gainsville, Florida
  - University of Maryland - Dental School, Baltimore, Maryland
  - Boston University Dental School, Boston, Massachusetts
  - University of Michigan Oral Health Research Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - State University of New York at Buffalo, Dental Medicine, Buffalo, New York
  - University of Pennsylvania Dental School, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Scaling and Root Planing + SHAM TX: Empty syringe + Scaling and root planing
- Scaling & Root Planing + Periocline Gel: Gel WITH Minocycline HCL 2.1% + Scaling & root planing
  minocycline HCl 2.1% : Minocycline HCl 2.1% gel as an adjunct to scaling and root planing. Dosing is by topical delivery into gingival pockets at baseline, 2 weeks, 4 weeks, 3 months and 6 months.
- Scaling and Root Planing + Vehicle: Gel WITHOUT 2.1% Minocycline HCl + Scaling and root planing
Period: Overall Study
Arm/Group | Scaling and Root Planing + SHAM TX | Scaling & Root Planing + Periocline Gel | Scaling and Root Planing + Vehicle
Started | 200 | 202 | 200
Completed | 171 | 172 | 174
Not Completed | 29 | 30 | 26

BASELINE CHARACTERISTICS:
Groups:
- Scaling and Root Planing + SHAM TX: sham treatment
  Scaling and root planing : scaling and root planing
- Scaling & Root Planing + Periocline Gel: Minocycline HCL 2.1%
  minocycline HCl 2.1% : Minocycline HCl 2.1% gel as an adjunct to scaling and root planing. Dosing is by topical delivery into gingival pockets at baseline, 2 weeks, 4 weeks, 3 months and 6 months.
- Scaling and Root Planing + Vehicle: Placebo
  Scaling and root planing : scaling and root planing
- Total: Total of all reporting groups
Arm/Group | Scaling and Root Planing + SHAM TX | Scaling & Root Planing + Periocline Gel | Scaling and Root Planing + Vehicle | Total
Number analyzed (Participants) | 200 | 202 | 200 | 602
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 193 | 196 | 198 | 587
  >=65 years | 7 | 6 | 2 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (11.5) | 49.2 (11.8) | 50.2 (12.0) | 49.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 108 | 93 | 300
  Male | 101 | 94 | 107 | 302
Region of Enrollment [Number; unit: participants]
  United States | 200 | 202 | 200 | 602

OUTCOME MEASURES:

1. Primary Outcome: Change in Pocket Depth.
Description: Average change of Pocket Depth at 9 months from baseline
Time Frame: baseline & 9 months
Population: Intent to treat
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Groups:
- Scaling and Root Planing + Periocline Gel: Minocycline HCL 2.1%
  minocycline HCl 2.1% : Minocycline HCl 2.1% gel as an adjunct to scaling and root planing. Dosing is by topical delivery into gingival pockets at baseline, 2 weeks, 4 weeks, 3 months and 6 months.
Arm/Group | Scaling and Root Planing + SHAM TX | Scaling and Root Planing + Periocline Gel | Scaling and Root Planing + Vehicle
Number analyzed (Participants) | 200 | 202 | 200
mm | -1.4 [-1.7 to -1.1] | -1.6 [-1.8 to -1.3] | -1.4 [-1.7 to -1.1]

ADVERSE EVENTS:
Arm/Group | Scaling and Root Planing + SHAM TX | Scaling & Root Planing + Periocline Gel | Scaling and Root Planing + Vehicle
Serious Adverse Events (participants affected / at risk) | 8/200 | 5/202 | 3/200
Other Adverse Events (participants affected / at risk) | 173/200 | 189/202 | 182/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scaling and Root Planing + SHAM TX (N=200) | Scaling & Root Planing + Periocline Gel (N=202) | Scaling and Root Planing + Vehicle (N=200)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Subject was involved in a motorcycle accident on 30 April 2006 and was hospitalized.
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Death (Social circumstances) | 0 (0) | 1 (1) | 0 (0) — Died in a car accident
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cellulitis and pulmonary embolism (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hysterectomy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction and fatigue (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Right knee replacement surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischemic attack (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Cellulitis of male organ external epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Hopsitalization for complications from Multiple Sclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain and injury (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cast (Social circumstances) | 0 (0) | 1 (1) | 0 (0) — Subject slipped on the ice in driveway. An x-ray showed a fracture of the left ankle. A cast was placed and subsequently replaced with a brace enabling the subject to walk without assistive devices.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scaling and Root Planing + SHAM TX (N=200) | Scaling & Root Planing + Periocline Gel (N=202) | Scaling and Root Planing + Vehicle (N=200)
Gastrointestinal disorders (Gastrointestinal disorders) | 138 (412) | 140 (430) | 134 (338) — Collected in a non-specific manner
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 71 (129) | 137 (485) | 138 (495) — Collected in a non-specific manner
Gerenal Disorders and adminstration site conditions (General disorders) | 30 (43) | 131 (141) | 109 (116) — Collected in a non-specific manner
Infections and infestations (Infections and infestations) | 44 (63) | 41 (51) | 40 (50) — Collected in a non-specific manner
Nervous system disorders (Nervous system disorders) | 16 (78) | 11 (16) | 16 (27) — Collected in a non-specific manner
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 12 (35) | 16 (23) | 11 (11) — Collected in a non-specific manner
Respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 27 (41) | 19 (30) | 25 (36) — Collected in a non-specific manner

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other